CLINICAL TRIAL: NCT04922177
Title: Computer-aided Design/Computer-aided Manufacturing for Mild to Moderate Molar Incisor Hypomineralization Treatment : a Pilot Study
Brief Title: Computer-aided Design/Computer-aided Manufacturing for Mild to Moderate Molar Incisor Hypomineralization Treatment
Acronym: MIhCFAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/19/0053
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor Hypomineralization; Direct restauration; Computer-aided design (CAD); Computer-aided manufacturing (CAM)
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM Group (Experimental): For the CAD/CAM group, an indirect ceramic restoration will be made using an optical impression.
  Interventions: Procedure: Indirect ceramic restoration
- Direct method Group (Active Comparator): For the direct method group, a restoration using a Glass Ionomer Cement will be performed.
  Interventions: Procedure: Direct restoration

INTERVENTIONS:
Procedure: Indirect ceramic restoration — Indirect ceramic restoration using an optical impression.
  Arms: CAD/CAM Group
Procedure: Direct restoration — Restoration using a Glass Ionomer Cement
  Arms: Direct method Group

SUMMARY:
Molar Incisor Hypomineralization (MIH) is a disease causing a structural defect in the enamel of permanent teeth. The treatment of these teeth consists of the removal of the affected part of the tooth and its reconstitution. Classically, the restoration is done with a resin in direct method. With the development of Computer-aided design (CAD) and Computer-aided manufacturing (CAM), it is possible to make a custom-made part to replace the affected part of the tooth. The main objective is to describe the effect of the 6-month management of CAD/CAM type restorations compared to direct restorations, performed in children aged 7 to 12 years with mild to moderate MIH on permanent molar teeth.

DETAILED DESCRIPTION:
Molar Incisor Hypomineralization (MIH) is a structural defect of the enamel affecting at least one of the first four permanent molars. The prevalence is high, ranging from 20% to 40% of children. The consequences of MIH are multiple, including pain during food intake or an increased risk for the development of carious disease. The current standard protocol for mild to moderate MIH is the use of direct restorations (Glass Cement Ionomer type). However, this therapy is not suitable due to frequent failures. In terms of longevity, indirect restorations are superior to direct restorations. CAD/CAM in dentistry offers the possibility of making these inlay/onlay type perennial coronary restorations. It is faster to implement and does not require a conventional impression.

ELIGIBILITY:
* inclusion criteria:

  1. Child from 7 to 12 years old presenting a mild to moderate HIN on at least one permanent first molar requiring reconstitution.
  2. Child presenting a state of anxiety compatible with the provision of oral care (score on the Venham scale modified by Veerkamp below 2).
  3. Child affiliated to or benefiting from a social security scheme.
  4. Free, informed and signed consent by the parent(s)/holder(s) of parental authority and the investigator (at the latest on the day of inclusion and before any examination required by the research).
  5. Oral consent of the child.
* Non-inclusion criteria:

  1. Child presenting an allergy or a history of allergy to one of the constituents of biomaterials
  2. Child with fluorosis
  3. Child with amelogenesis imperfecta
  4. Child with pacemaker (contraindication to CAD/CAM)

     -

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Treatment effect | 6 months
  The effect of the management of the MIH will be assessed by the occurrence of failure. Failure will be diagnosed from the degree of demineralisation measured, by laser fluorescence at the peripheral tooth/restoration joint. The values collected range from 0 to 99 and are categorised into 3 situations :
  * From 0 to 12: situation without demineralization, tight seal.
  * From 13 to 24: start of demineralization
  * ≥ 25: therapeutic failure, non-watertight seal, restoration to be redone without delay.

SECONDARY OUTCOMES:
Failure | 3 months
  Failure diagnosed according to the degree of demineralisation measured, every 3 months following the restoration, by laser fluorescence at the peripheral tooth/restoration joint.
Failure | 12 months
  Failure diagnosed according to the degree of demineralisation measured, every 12 months following the restoration, by laser fluorescence at the peripheral tooth/restoration joint.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu MARTY, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University hospital of Toulouse, Toulouse, France